CLINICAL TRIAL: NCT05957666
Title: Comparison of Oral Versus Vaginal Misoprostol for Labour Induction at Term
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Tayyiba Wasim, Professor Obstetrics and Gynaecology, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB/2023/1129/SIMS
Record Dates: First submitted 2023-07-15; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Induction of Labour With Misoprostol
Keywords: induction of labour; misoprostol
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: Total 176 patient included in this study.Patients will be randomised by envelop method to recieve either oral or vaginal misoprostol in a dose of 50microgram.
Who Masked: Participant, Investigator
Masking Description: patients will either recieve oral or vaginal misoprostol by envelope method ina dose of 50microgram.Total of 176 envelopes are placed in a concealed box.Neither the doctor nor the patient knows.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oral misoprostol (Experimental): oral misoprostol will be given in a dose of 50microgram and repeated after 6 hours if required.Maximum 2 doses will be given
  Interventions: Drug: Misoprostol Oral Tablet
- vaginal misoprostol (Active Comparator): vaginal misoprostol will be given in a dose of 50 microgram and repeated after 6 hours if required.Maximum 2 doses will be given
  Interventions: Drug: vaginal misoprostol

INTERVENTIONS:
Drug: Misoprostol Oral Tablet — oral misoprostol 50 microgram repeated after 6 hours if required
  Other Names: cytotec
  Arms: oral misoprostol
Drug: vaginal misoprostol — vaginal misoprostol 50 microgram repeated after 6 hours if required
  Other Names: cytotec
  Arms: vaginal misoprostol

SUMMARY:
A randomised control trial to compare oral and vaginal misoprostol for induction of labour in term patients.The objective is to determine whether use of standardised vaginal misoprostol regimen will result in decreased cesaerean section rate among women with bishop score of lessthan or equal to 6 who require induction of labpour at term compared to oral misoprostol regimen.

DETAILED DESCRIPTION:
The objective of study is to determine whether the use of standardised vaginal misoprostol regimen will result in decreased cesaerean section rate among women with bishop score of less than or equal to 6 who require induction of labour at term compared to oral misoprostol regimen.It is a randomised control trial conducted in department of obs and gynae unit 1 from june 2023.

Total 176 patients are included in this study and they will be randomised by envelope method to recieve either oral or vaginal misoprostol in a dose of 50microgram.In both groupds dose will be repeated after 6 hours if required.Maximum 2 doses will be given.patients will be monitored for uterine contractions and fetal hearts.Vaginal examination will be done at 4hours and 8 hours following misoprostol dose or earlier if patient complains of leaking and labour pains.Membranes will be ruptured once cervical dilatation is greater than 3cm.in absence of adequate uterine contractions oxytocin infusion will be started.Fetal hearts will be monitored every 30 minutes from time of induction.Progress of labour will be assessed through partogram.

ELIGIBILITY:
Inclusion Criteria:

Cephalic presentation Prelabour rupture of membranes Singleton pregnancies reaching 41 weeks G1 to G4 Bishop score of less than or equal to 6 Medical disorders(GDM,PIH) -

Exclusion Criteria:

Previous uterine scar Antepartum hemorrhage Cephalopelvic disproportion Multiple gestation Multiparity Oligohydramnios/polyhydramnios IUGR Severe systemic illness like pre eclampsia,eclampsia,cardiac,hepatic,renal disease PPROM

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-12-16 (Estimated); Study Completion 2023-12-16 (Estimated)

PRIMARY OUTCOMES:
vaginal birth | vaginal birth within 24 hours of admission
  vaginal birth within 24 hours of admission with 2 doses of misoprostol given 6 hours apart

SECONDARY OUTCOMES:
cesaerean section | within 24 hours
  cesaerean section if patient doesnt go in labour despite 2 doses or fetal distress occurs
induction to delivery interval | within 24 hours
  measured from 1st dose till delivery of patient
fetal distress | within 24 hours
  fetal distress measured by non reactive CTG or meconium stained amniotic fluid
uterine hyperstimulation | more than 10 cotractions in every 10 minutes
  more than 5 contractions in every 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Services Institute Of Medical Sciences, Lahore, Punjab Province, Pakistan